CLINICAL TRIAL: NCT02894502
Title: MOTIVATional intErviewing to Improve Self-care in Heart Failure Patients (MOTIVATE-HF): Study Protocol of a Three-arm Multicenter Randomized Controlled Trial
Brief Title: MOTIVATional intErviewing to Improve Self-care in Heart Failure Patients
Acronym: MOTIVATE-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rome Tor Vergata (Other)
Collaborators: Center of Excellence for Nursing Scholarship (Other)
Responsible Party: Principal Investigator, Ercole Vellone, Assistant Professor, University of Rome Tor Vergata
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 121/13
Record Dates: First submitted 2016-08-26; First posted 2016-09-09 (Estimated); Results first posted 2021-02-24 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-02

CONDITIONS: Heart Failure
Keywords: Self-care; Motivational interviewing; Heart failure; Caregivers
MeSH Terms: conditions — Heart Failure | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Motivational interviewing only for patients (Experimental): In this arm the interventions will be delivered only to patients
  Interventions: Behavioral: Motivational interviewing
- Motivational interviewing to patients and caregivers (Experimental): In this arm the interventions will be delivered both to patients and caregivers
  Interventions: Behavioral: Motivational interviewing
- Control group (No Intervention): This Group will receive the usual care

INTERVENTIONS:
Behavioral: Motivational interviewing — The intervention will consist of a brief session of motivational interviewing (MI) performed by a trained nurse. During MI, the interventionist will address one or two aspects of self-care that the participants want to address. After this first intervention, the same interventionist will contact the participant by telephone to improve the first intervention and provide further support as needed. These telephone contact will be done three times at two week intervals following the first intervention (for a total of two months). Patients and caregivers that receive the intervention also will be given informational material on HF management that is consistent with international guidelines.
  Arms: Motivational interviewing only for patients; Motivational interviewing to patients and caregivers

SUMMARY:
The aims of this study will be to evaluate the effect of motivational interviewing (MI) to improve self-care in heart failure (HF) patients and caregiver contributions to HF self-care. Also this study will evaluate the effect of MI on the following secondary outcomes: In HF patients: HF somatic symptom perception, generic and specific quality of life, anxiety and depression, sleep quality, mutuality with caregiver, hospitalizations, use of emergency services, and mortality; In caregivers: generic quality of life, anxiety and depression, mutuality with patient, preparedness, social support and sleep quality.

ELIGIBILITY:
Inclusion criteria:

Diagnosis of HF (for patient), New York Heart Association (NYHA) functional class II- IV (for patient), Inadequate self-care assessed with the Self-Care Heart Failure Index (for patient), Being the informal caregiver of the patients (for caregiver).

Exclusion criteria:

Severe cognitive impairment evaluated with the Six-item screener (for patient), Acute coronary syndrome during the last three months (for patient), Living in a residential settings (e.g., nursing home) (for patient), Patients not willing to participate in the study (for caregiver).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Actual)
Dates: Start 2014-06; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rome Tor Vergata, Rome, Italy

IPD SHARING:
Plan to Share IPD: Yes
In case there will be the possibility to share the data, this will be done after data de-identification

REFERENCES:
- [Background] Vellone E, Paturzo M, D'Agostino F, Petruzzo A, Masci S, Ausili D, Rebora P, Alvaro R, Riegel B. MOTIVATional intErviewing to improve self-care in Heart Failure patients (MOTIVATE-HF): Study protocol of a three-arm multicenter randomized controlled trial. Contemp Clin Trials. 2017 Apr;55:34-38. doi: 10.1016/j.cct.2017.02.003. Epub 2017 Feb 7. PMID 28185994
- [Result] Vellone E, Rebora P, Ausili D, Zeffiro V, Pucciarelli G, Caggianelli G, Masci S, Alvaro R, Riegel B. Motivational interviewing to improve self-care in heart failure patients (MOTIVATE-HF): a randomized controlled trial. ESC Heart Fail. 2020 Jun;7(3):1309-1318. doi: 10.1002/ehf2.12733. Epub 2020 Apr 28. PMID 32343483
- [Derived] Iovino P, Dollaku H, Alvaro R, Pucciarelli G, Rasero L, Macchi C, Liuzzi P, Riegel B, Vellone E. Sleep quality patterns in patients with heart failure: a person-centred latent class analysis from a secondary analysis of the MOTIVATE-HF trial. BMJ Open. 2025 Aug 8;15(8):e101950. doi: 10.1136/bmjopen-2025-101950. PMID 40780724
- [Derived] Iovino P, Dollaku H, Rasero L, Uchmanowicz I, Alvaro R, Pucciarelli G, Vellone E. Psychometric Testing of the Kansas City Cardiomyopathy Questionnaire 12 in A European Population. J Cardiovasc Nurs. 2025 Feb 27;40(6):E374-82. doi: 10.1097/JCN.0000000000001187. Online ahead of print. PMID 40013908
- [Derived] Caggianelli G, Alivernini F, Chirico A, Iovino P, Lucidi F, Uchmanowicz I, Rasero L, Alvaro R, Vellone E. The relationship between caregiver contribution to self-care and patient quality of life in heart failure: A longitudinal mediation analysis. PLoS One. 2024 Mar 12;19(3):e0300101. doi: 10.1371/journal.pone.0300101. eCollection 2024. PMID 38470867
- [Derived] Locatelli G, Iovino P, Jurgens CY, Alvaro R, Uchmanowicz I, Rasero L, Riegel B, Vellone E. The Influence of Caregiver Contribution to Self-care on Symptom Burden in Patients With Heart Failure and the Mediating Role of Patient Self-care: A Longitudinal Mediation Analysis. J Cardiovasc Nurs. 2024 May-Jun 01;39(3):255-265. doi: 10.1097/JCN.0000000000001024. Epub 2023 Aug 8. PMID 37550831
- [Derived] Locatelli G, Rebora P, Occhino G, Ausili D, Riegel B, Cammarano A, Uchmanowicz I, Alvaro R, Vellone E, Zeffiro V. The Impact of an Intervention to Improve Caregiver Contribution to Heart Failure Self-care on Caregiver Anxiety, Depression, Quality of Life, and Sleep. J Cardiovasc Nurs. 2023 May 18;38(4):361-9. doi: 10.1097/JCN.0000000000000998. Online ahead of print. PMID 37204336
- [Derived] Spedale V, Fabrizi D, Rebora P, Luciani M, Alvaro R, Vellone E, Riegel B, Ausili D. The Association Between Self-reported Sleep Quality and Self-care in Adults With Heart Failure: A Cross-sectional Study. J Cardiovasc Nurs. 2023 May-Jun 01;38(3):E98-E109. doi: 10.1097/JCN.0000000000000929. Epub 2022 May 31. PMID 37027137
- [Derived] Locatelli G, Zeffiro V, Occhino G, Rebora P, Caggianelli G, Ausili D, Alvaro R, Riegel B, Vellone E. Effectiveness of Motivational Interviewing on contribution to self-care, self-efficacy, and preparedness in caregivers of patients with heart failure: a secondary outcome analysis of the MOTIVATE-HF randomized controlled trial. Eur J Cardiovasc Nurs. 2022 Nov 23;21(8):801-811. doi: 10.1093/eurjcn/zvac013. PMID 35290454
- [Derived] Caggianelli G, Iovino P, Rebora P, Occhino G, Zeffiro V, Locatelli G, Ausili D, Alvaro R, Riegel B, Vellone E. A Motivational Interviewing Intervention Improves Physical Symptoms in Patients with Heart Failure: A Secondary Outcome Analysis of the Motivate-HF Randomized Controlled Trial. J Pain Symptom Manage. 2022 Feb;63(2):221-229.e1. doi: 10.1016/j.jpainsymman.2021.09.006. Epub 2021 Sep 25. PMID 34571194
- [Derived] Rebora P, Spedale V, Occhino G, Luciani M, Alvaro R, Vellone E, Riegel B, Ausili D. Effectiveness of motivational interviewing on anxiety, depression, sleep quality and quality of life in heart failure patients: secondary analysis of the MOTIVATE-HF randomized controlled trial. Qual Life Res. 2021 Jul;30(7):1939-1949. doi: 10.1007/s11136-021-02788-3. Epub 2021 Feb 22. PMID 33616815

RESULTS

PARTICIPANT FLOW:
Period: Baseline
Arm/Group | Motivational Interviewing Only for Patients | Motivational Interviewing to Patients and Caregivers | Control Group
Started | 155 | 177 | 178
Completed | 128 | 145 | 133
Not Completed | 27 | 32 | 45
Not completed — Withdrawal by Subject | 24 | 31 | 36
Not completed — Death | 3 | 1 | 9
Period: First Follow up
Arm/Group | Motivational Interviewing Only for Patients | Motivational Interviewing to Patients and Caregivers | Control Group
Started | 128 | 145 | 133
Completed | 94 | 114 | 93
Not Completed | 34 | 31 | 40
Not completed — Withdrawal by Subject | 32 | 29 | 37
Not completed — Death | 2 | 2 | 3
Period: Second Follow up
Arm/Group | Motivational Interviewing Only for Patients | Motivational Interviewing to Patients and Caregivers | Control Group
Started | 94 | 114 | 93
Completed | 79 | 96 | 79
Not Completed | 15 | 18 | 14
Not completed — Withdrawal by Subject | 13 | 15 | 13
Not completed — Death | 2 | 3 | 1
Period: Third Follow up
Arm/Group | Motivational Interviewing Only for Patients | Motivational Interviewing to Patients and Caregivers | Control Group
Started | 79 | 96 | 79
Completed | 73 | 89 | 76
Not Completed | 6 | 7 | 3
Not completed — Withdrawal by Subject | 5 | 6 | 3
Not completed — Death | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Motivational Interviewing Only for Patients | Motivational Interviewing to Patients and Caregivers | Control Group | Total
Number analyzed (Participants) | 155 | 177 | 178 | 510
Age, Categorical [Count of Participants; unit: Participants] — Population: In the "Motivational interviewing only for patients" and in the "Control group" Arms we have missing data.
  Participants
    number analyzed (Participants) | 154 | 177 | 177 | 508
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 35 | 45 | 47 | 127
    >=65 years | 119 | 132 | 130 | 381
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: In the first and in the third arm we have missing data
  Years
    number analyzed (Participants) | 154 | 177 | 177 | 508
    (all) | 72.19 (12.29) | 72.45 (10.79) | 72.45 (13.66) | 72.37 (12.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 70 | 69 | 214
  Male | 80 | 107 | 109 | 296
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 155 | 177 | 178 | 510
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Self-Care of Heart Failure Index [Mean (Standard Deviation); unit: units on a scale] — Score of the Self-Care Maintenance Scale of the Self-Care of Heart Failure Index (SCHFI) (primary endpoint). The SCHFI has three scales: Self-Care Maintenance, Self-Care Management and Self-Care Confidence. Each scale has a score from 0 to 100 with higher score meaning better self-care. Self-Care is considered adequate when patients have a score at each scale of 70 at least.
  units on a scale | 45.72 (15.23) | 45.98 (16.35) | 44.98 (14.61) | 45.55 (15.39)
Heart Failure Somatic Perception Scale [Mean (Standard Deviation); unit: units on a scale] — The Heart Failure Somatic Perception Scale has a score between 0 and 90 with higher scores meaning more discomfort caused by heart failure symptoms
  units on a scale | 30.55 (18.20) | 30.18 (18.25) | 31.83 (18.95) | 30.87 (18.46)
SF-12 (Physical Component Summary) [Mean (Standard Deviation); unit: units on a scale] — The SF-12 (Physical Component Summary) measures the physical aspects of health-related quality of life. The score ranges between 0 and 100 with higher score indicating better quality of life.
  units on a scale | 36.01 (10.35) | 35.01 (9.16) | 35.42 (9.30) | 35.46 (9.57)

OUTCOME MEASURES:

1. Primary Outcome: Self-care Maintenance in Patients
Description: Self-care in HF patients will be measured with the Self-Care of HF Index V.6.2. Since this instrument has three separate scales, we considered as a primary outcome the score of the Self-care Maintenance scale. The Self-Care Maintenance scale has a score between 0 and 100 with higher score meaning better self-care. Self-Care Maintenance is considered adequate when the score is at least 70.
Time Frame: 3 months from the intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Motivational Interviewing Only for Patients | Motivational Interviewing to Patients and Caregivers | Control Group
Number analyzed (Participants) | 128 | 145 | 133
score on a scale | 52.36 (22.67) | 54.23 (20.36) | 49.63 (17.49)

2. Secondary Outcome: Burden of HF Symptoms in Patients
Description: Burden of HF symptoms will be measured with the Heart Failure Somatic Perception Scale (HFSPS). The HFSPS has a range score between 0 and 90; the higher the score, the higher the burden of symptoms caused by heart failure.
Time Frame: 3, 6, 9 and 12 months from the intervention
Population: Patients with heart failure
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Motivational Interviewing Only for Patients: In this Arm, motivational interviewing will be provided only to patients
- Motivational Interviewing for Patients and Caregivers: In this Arm, motivational interviewing will be provided to patients and caregivers
- Control Group: This Arm will receive the standard of care
Arm/Group | Motivational Interviewing Only for Patients | Motivational Interviewing for Patients and Caregivers | Control Group
Number analyzed (Participants) | 73 | 89 | 76
score on a scale | 24 (16.5) | 17.4 (18.8) | 22.5 (21.7)

3. Secondary Outcome: Patient and Caregiver Generic Physical and Mental Quality of Life
Description: Patient and caregiver generic physical and mental quality of life will be assessed with the Short Form 12 (SF-12).
Time Frame: 3, 6, 9 and 12 months from the intervention
Reporting Status: Not Posted

4. Secondary Outcome: Patient and Caregiver Anxiety and Depression
Description: Patient and caregiver anxiety and depression will be evaluated with the Hospital Anxiety and Depression Scale
Time Frame: 3, 6, 9 and 12 months from the intervention
Reporting Status: Not Posted

5. Secondary Outcome: Patient HF Specific Quality of Life
Description: Patient HF specific quality of life will be evaluated with the Kansas City Cardiomyopathy Questionnaire
Time Frame: 3, 6, 9 and 12 months from the intervention
Reporting Status: Not Posted

6. Secondary Outcome: Patient and Caregiver Quality of Nocturnal Sleep
Description: We will use the Pittsburgh Sleep Quality Index
Time Frame: 3, 6, 9 and 12 months from the intervention
Reporting Status: Not Posted

7. Secondary Outcome: Patient and Caregiver Mutuality
Description: We will use the Mutuality Scale
Time Frame: 3, 6, 9 and 12 months from the intervention
Reporting Status: Not Posted

8. Secondary Outcome: Caregiver Preparedness
Description: Caregiver Preparedness will be evaluated with the Caregiver Preparedness Scale
Time Frame: 3, 6, 9 and 12 months from the intervention
Reporting Status: Not Posted

9. Secondary Outcome: Caregiver Perceived Social Support
Description: We will use the Multidimensional Scale of Perceived Social Support Scale
Time Frame: 3, 6, 9 and 12 months from the intervention
Reporting Status: Not Posted

10. Secondary Outcome: Patient Hospitalizations
Description: The number of patient hospitalizations will be measured asking the caregiver how many time the patient was hospitalized from at 3, 6, 9 and 12 months from the intervention.
Time Frame: 3, 6, 9 and 12 months from the intervention
Reporting Status: Not Posted

11. Secondary Outcome: Use of Emergency Services
Description: How many times the patient has used the emergency services will be evaluated by asking the caregiver how many time the patient used after 3, 6, 9 and 12 months from the intervention.
Time Frame: 3, 6, 9 and 12 months from the intervention
Reporting Status: Not Posted

12. Secondary Outcome: Death
Description: Death rates will be evaluated in the three arms of the study by caregiver interview at 3, 6, 9 and 12 months from the intervention.
Time Frame: 3, 6, 9 and 12 months from the intervention
Population: The above participants were those who were randomized initially in the three arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Interviewing Only for Patients | Motivational Interviewing to Patients and Caregivers | Control Group
Number analyzed (Participants) | 155 | 177 | 178
Participants
  3 month follow-up: Overall Number of Participants Analyzed | 128 | 145 | 133
  3 month follow-up: Number of Deaths | 3 | 1 | 9
  3 month follow-up: Number of refusals to continue the study | 24 | 31 | 36
  6 month follow-up: Overall Number of Participants Analyzed | 94 | 114 | 93
  6 month follow-up: Number of Deaths | 5 | 3 | 12
  6 month follow-up: Number of refusals to continue the study | 56 | 60 | 73
  9 month follow-up: Overall Number of Participants Analyzed | 79 | 96 | 79
  9 month follow-up: Number of Deaths | 7 | 6 | 13
  9 month follow-up: Number of refusals to continue the study | 69 | 75 | 86
  12 month follow-up: Overall Number of Participants Analyzed | 73 | 89 | 76
  12 month follow-up: Number of Deaths | 8 | 7 | 13
  12 month follow-up: Number of refusals to continue the study | 74 | 81 | 89

ADVERSE EVENTS:
Time Frame: one year
Description: In this study we considered only all-cause mortality.
Arm/Group | Motivational Interviewing Only for Patients | Motivational Interviewing to Patients and Caregivers | Control Group
All-Cause Mortality (participants affected / at risk) | 8/155 | 7/177 | 13/178
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-09): https://cdn.clinicaltrials.gov/large-docs/02/NCT02894502/Prot_SAP_000.pdf